CLINICAL TRIAL: NCT02832154
Title: Enhancing Management of Patient Reported Outcomes With Emotion Regulation (EMPOWER)
Brief Title: Internet-Delivered Positive Affect Program in Managing Emotion in Young Adult Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00037913; NCI-2016-00647 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCCWFU 99516 (Other: Comprehensive Cancer Center of Wake Forest University); P30CA012197 (NIH); R01MH084723 (NIH)
Record Dates: First submitted 2016-05-20; First posted 2016-07-14 (Estimated); Results first posted 2020-07-16 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Cancer Survivor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive Care (Experimental): Patients complete an initial online questionnaire lasting about 25-30 minutes. Patients complete an internet-delivered PA program during weeks 3-8. Each week consists of didactic material and 20-30 minutes of daily online exercises.
  Interventions: Other: Internet-Based Intervention; Procedure: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Internet-Based Intervention — Complete online PA program
Procedure: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This pilot clinical trial studies how well an internet-delivered positive affect (PA) intervention works in managing emotion in young adult cancer survivors. An internet-delivered PA intervention may teach younger cancer survivors healthy coping skills and help doctors to learn more about what effects mood may have on the health and well-being of young adults with cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To adapt an individualized positive affect intervention that was developed for newly diagnosed HIV patients to use with young adult cancer survivors.

II. To pilot test the positive affect intervention with young adult cancer survivors to determine its feasibility and acceptability.

SECONDARY OBJECTIVES:

I. To describe health related quality of life, psychological well-being, daily emotion reports, and health behaviors in young adult cancer survivors.

OUTLINE:

Patients complete an initial online questionnaire lasting about 25-30 minutes. Patients complete an internet-delivered PA program during weeks 3-8. Each week consists of didactic material and 20-30 minutes of daily online exercises.

After completion of study, patients are followed up at 1 and 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Able to read and understand English
* Past history of a cancer diagnosis (excluding basal cell skin carcinoma)
* 18 to 39 years of age at diagnosis
* Within 0-5 years post-active treatment
* Wireless internet connection or a home computer that is connected to the internet

Exclusion Criteria:

* Evidence of a cancer recurrence
* History of multiple primary cancers
* Currently receiving palliative or hospice care
* Significant psychiatric history

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2017-04-21 (Actual); Primary Completion 2019-04-23 (Actual); Study Completion 2020-04-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Salsman, Principal Investigator — Wake Forest University Health Sciences
Locations (2):
- United States (2):
  - Northwestern University, Chicago, Illinois
  - Comprehensive Cancer Center of Wake Forest University, Winston-Salem, North Carolina

REFERENCES:
- [Derived] Salsman JM, McLouth LE, Tooze JA, Little-Greene D, Cohn M, Kehoe MS, Moskowitz JT. An eHealth, Positive Emotion Skills Intervention for Enhancing Psychological Well-Being in Young Adult Cancer Survivors: Results from a Multi-Site, Pilot Feasibility Trial. Int J Behav Med. 2023 Oct;30(5):639-650. doi: 10.1007/s12529-023-10162-5. Epub 2023 Mar 8. PMID 36890329
- [Derived] Salsman JM, McLouth LE, Cohn M, Tooze JA, Sorkin M, Moskowitz JT. A Web-Based, Positive Emotion Skills Intervention for Enhancing Posttreatment Psychological Well-Being in Young Adult Cancer Survivors (EMPOWER): Protocol for a Single-Arm Feasibility Trial. JMIR Res Protoc. 2020 May 28;9(5):e17078. doi: 10.2196/17078. PMID 32463014

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Supportive Care
Started | 43
Completed | 43
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Supportive Care
Number analyzed (Participants) | 43
Age, Continuous [Mean (Standard Deviation); unit: Years] | 30.37 (6.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 40
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 35
  More than one race | 2
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 43

OUTCOME MEASURES:

1. Primary Outcome: Acceptability - Mean Value
Description: Quantitative measures and interview will be used to quantify acceptability. The mean of participants responding affirmatively to the highest two responses from an intervention evaluation phone interview script created by investigators will be combined and exact 95% confidence intervals (CIs) will be calculated for these estimates. Participants were asked the following questions: On a scale of 0 to 10, with 0 being definitely not to 10 being definitely yes, to what extent would you recommend these skills to a friend? and To what extent would you recommend this intervention to someone newly diagnosed with cancer?
Time Frame: At 12 weeks
Population: Only 26 participants out of the 43 were analyzed for acceptability for this outcome.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Supportive Care
Number analyzed (Participants) | 26
score on a scale | 8.81 [8.27 to 9.34]

2. Primary Outcome: Acceptability - Proportion Value
Description: Quantitative measures and interview will be used to quantify acceptability. The proportion of participants responding affirmatively to the highest two responses from an intervention evaluation phone interview script created by investigators will be combined and exact 95% confidence intervals (CIs) will be calculated for these estimates. Responding affirmatively means a score of 9 or 10 on the scale of 0-10, so the proportion responding affirmatively is the proportion of patients who responded with a 9 or 10 to those questions. Participants were asked the following questions: On a scale of 0 to 10, with 0 being definitely not to 10 being definitely yes, to what extent would you recommend these skills to a friend? and To what extent would you recommend this intervention to someone newly diagnosed with cancer?
Time Frame: At 12 weeks
Population: Only 26 participants out of the 43 were analyzed for acceptability for this outcome.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Supportive Care
Number analyzed (Participants) | 26
proportion of participants | 0.58 [0.37 to 0.77]

3. Primary Outcome: Accrual
Description: Accrual will be estimated as the number of patients accrued divided by the number of months of accrual. A 95% confidence interval for the monthly accrual rate will be calculated based on the Poisson distribution.
Time Frame: Up to 19 months
Measure: Mean (95% Confidence Interval); unit: participants per month
Arm/Group | Supportive Care
Number analyzed (Participants) | 43
participants per month | 1.63 [1.18 to 2.19]

4. Primary Outcome: Adherence - Proportion of Completed Interventions (Mean Value)
Description: Adherence to the intervention will be calculated as the number of intervention sessions completed. Investigators will calculate and report the mean adherence across all individuals who completed three or more sessions.
Time Frame: At 12 weeks
Measure: Mean (Standard Deviation); unit: completed interventions
Arm/Group | Supportive Care
Number analyzed (Participants) | 43
completed interventions | 3.30 (2.20)

5. Primary Outcome: Adherence - Proportion of Completed Interventions (Proportion Value)
Description: Adherence to the intervention will be calculated as the number of intervention sessions completed. Investigators will calculate and report the proportion of patients who completed three or more sessions.
Time Frame: At 12 weeks
Measure: Mean (Standard Deviation); unit: complete interventions
Arm/Group | Supportive Care
Number analyzed (Participants) | 43
complete interventions | 0.63 (0.48)

6. Primary Outcome: Number of Patients Who Refused to Participate
Description: The refusal rate will be estimated as the number of patients who refuse to participate divided by the number eligible.
Time Frame: At 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Supportive Care
Number analyzed (Participants) | 43
Participants | 27

7. Primary Outcome: Number of Patient Provided Data at 8 Weeks - Retention
Description: Retention will be defined as the proportion of patients who provide 8 week data. Patients who discontinue the intervention (refuse phone calls) but complete the outcome assessments will be counted in the numerator for calculating retention. Retention estimates will be calculated overall and by site
Time Frame: At 8 week
Measure: Count of Participants; unit: Participants
Arm/Group | Supportive Care
Number analyzed (Participants) | 43
Participants | 27

8. Primary Outcome: Adherence - Number of Completed Exercises
Description: Adherence to the intervention will be calculated as the frequency of completing exercises. Investigators will calculate and report the mean adherence across all individuals as well as the proportion of patients who completed three or more sessions.
Time Frame: At 12 weeks
Measure: Mean (Standard Deviation); unit: completed exercises
Arm/Group | Supportive Care
Number analyzed (Participants) | 43
completed exercises | 5.07 (3.43)

9. Primary Outcome: Number of Website Visits
Description: Adherence to the intervention will be calculated as the number of website visits. Investigators will calculate and report the mean adherence across all individuals as well as the proportion of patients who completed three or more sessions.
Time Frame: At 12 weeks
Measure: Mean (Standard Deviation); unit: website visits
Arm/Group | Supportive Care
Number analyzed (Participants) | 43
website visits | 15.35 (12.85)

10. Primary Outcome: Number of Patients Provided Data at 12 Weeks - Retention
Description: Retention will be defined as the number of patients who provide 12 week data. Patients who discontinue the intervention (refuse phone calls) but complete the outcome assessments will be counted in the numerator for calculating retention.
Time Frame: At 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Supportive Care
Number analyzed (Participants) | 43
Participants | 27

ADVERSE EVENTS:
Time Frame: Up to 19 months
Description: Adverse events were not monitored/assessed for this trial.
Arm/Group | Supportive Care
All-Cause Mortality (participants affected / at risk) | 0/43
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-12-29): https://cdn.clinicaltrials.gov/large-docs/54/NCT02832154/Prot_SAP_000.pdf
  • Informed Consent Form (2018-12-17): https://cdn.clinicaltrials.gov/large-docs/54/NCT02832154/ICF_001.pdf